CLINICAL TRIAL: NCT04397068
Title: Vergelijking Van de Postoperatieve Effectieve Lenspositie (ELP) Bij patiënten Gepland Voor Een Electieve Phacovitrectomie-ingreep (Phaco-VTX) Aan één Oog en Enkel Een Lensingreep Phaco Aan Het Andere Oog
Brief Title: Compare ELP in Patients With Elective Phaco-VTX Surgery in One Eye and a Single Lens Phaco Surgery on the Other Eye
Acronym: ELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. Peter Stalmans, Phd, MD, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S58904
Record Dates: First submitted 2016-03-14; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Macular Pucker
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- macular pucker wherefore vitrectomy (Other): one eye phaco-vitrectomy and other eye only phaco. No other involvement of drug or device. Standard of care procedure
  Interventions: Procedure: phaco-vitrectomy

INTERVENTIONS:
Procedure: phaco-vitrectomy — phaco-vitrectomy. No other involvement drug or device. Standard of care procedure

SUMMARY:
The aim of the study is to gain more insight into the potential impact of a vitrectomy (removal of the vitreous) on postoperative effective position of the intraocular lens (IOL). Moreover, this study can provide very useful information for the optimal lens calculation in patients undergoing lens extraction with IOL implantation (whether or not combined with a vitrectomy) should undergo.

DETAILED DESCRIPTION:
* Comparison ELP post phaco VTX (pucker / floaters) versus post phaco and use this information to develop a customized IOL calculation for eyes undergoing phacoVTX.
* Evidence for recording lens thickness (LT) parameter in the IOL strength calculation in KWS (in the calculation of the ELP in the light of the Olsen formula, using the C-constant) in order to be able to make an even more accurate prediction of the post-operative diopter target of the patient.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 yrs
* macular pucker wherefore vitrectomy is necessary

Exclusion Criteria:

* macular pathology other than macular pucker
* Corneal pathology
* Other ocular pathology that could affect the biometrics or ELP
* Previous vitrectomy in one of the eyes

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Compare if ELP is different or the same at phaco or phaco-vitrectomy | 6 - 8 weeks
  Anterior chamber depth measured using IOL master.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No